CLINICAL TRIAL: NCT04865640
Title: Clinical Validation Study for Noninvasive Cardiopulmonary Management Device.
Status: Completed | Type: Observational
Sponsor: Analog Device, Inc. (Other)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.1, 15Oct2020
Record Dates: First submitted 2021-04-23; First posted 2021-04-29 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Cardiopulmonary Disease
MeSH Terms: conditions — Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy Cohort: The target population for this cohort is healthy adult volunteers who do not have preexisting heart or lung conditions or illness. The goal is to recruit a participant population with a range of body types and BMIs and an approximately even split of genders.
  Interventions: Diagnostic Test: Noninterventional and noninvasive
- Pathologic Cohort: The target population for this cohort is adult patients who have been diagnosed with cardiopulmonary conditions. These can include chronic pulmonary conditions, chronic cardiac conditions, and those who are taking diuretic medications, living with heart failure, Chronic Obstructive Pulmonary Disorder (COPD), or recovering from coronary-artery disease-related events. The goal is to recruit a participant population with a range of body types and BMIs and an approximately even split of genders as well as conditions outlined above (e.g. at least 5 each of COPD, HF, recovering from a coronary artery disease-related event, and taking diuretic medication)
  Interventions: Diagnostic Test: Noninterventional and noninvasive

INTERVENTIONS:
Diagnostic Test: Noninterventional and noninvasive — The ADI At-Home CPM (Cardiopulmonary Management) System is intended for adults undergoing monitoring for cardiopulmonary conditions under the direction of a licensed medical professional to measure, record, and periodically transmit physiological data.

SUMMARY:
The ADI At-Home CPM (Cardiopulmonary Management) System is a non-invasive device that measures and trends a variety of biological parameters.

This study will be conducted as a prospective non-randomized study with two study arms/cohorts - one of healthy adult patients, one of pathologic patients who fit into the intended use population of the CPM System.

ELIGIBILITY:
Inclusion Criteria:

I. Healthy Cohort:

1. Adults over the age of 18 and who are willing and able to give informed consent.
2. Willing to participate in all activities related to this study, including trimming chest hair and wearing a reference device and the CPM wearable device.
3. Volunteers of any race, any gender
4. Range of physiques
5. Healthy

II. Pathologic Cohort

1. Adults over the age of 21 and who are willing and able to give informed consent
2. Willing to participate in all activities related to this study, including wearing a capnography device, thoracic impedance reference device, and the CPM wearable device.
3. Those who:

   1. Are taking diuretic medications
   2. Are living with heart failure
   3. Have chronic obstructive pulmonary disorder (COPD)
   4. Are recovering from a coronary-artery disease-related event.
4. Volunteers of any race, any gender-Range of physiques.

Exclusion Criteria:

I. Healthy Cohort

1. Injury or skin disturbance in the area of the test device
2. Pregnant
3. Currently smokes cigarettes
4. Has known respiratory conditions such as:

   1. Flu
   2. Pneumonia/bronchitis
   3. Shortness of breath/respiratory distress
   4. Respiratory or lung surgery
   5. Emphysema, COPD, lung disease
5. Has self-reported heart or cardiovascular conditions such as chest pain, AFib, CHF, cardiomyopathy, or other conditions that could interfere with cardiopulmonary function
6. Has other self-reported health conditions that could interfere with the breathing patterns and exercises detailed in the protocol (including wearing a capnography mask)

II. Pathologic Cohort:

1. Under the age of 21
2. Cognitive or physical impairment sufficient enough to interfere with informed consent or successful completion of the protocol.
3. Injury or skin disturbance in the area of the test device.
4. Pregnant.
5. Have life-threatening arrhythmias which require hospital admission and constant monitoring.
6. Has other self-reported health conditions that could interfere with wearing a capnography mask.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Cohort The target population for this cohort is healthy adult volunteers who do not have preexisting heart or lung conditions or illness. The goal is to recruit a participant population with a range of body types and BMIs and an approximately even split of genders.
  Pathologic Cohort The target population for this cohort is adult patients who have been diagnosed with cardiopulmonary conditions. These can include chronic pulmonary conditions, chronic cardiac conditions, and those who are taking diuretic medications, living with heart failure, Chronic Obstructive Pulmonary Disorder (COPD), or recovering from coronary-artery disease related events. The goal is to recruit a participant population with a range of body types and BMIs and an approximately even split of genders as well as conditions outlined above (e.g. at least 5 each of COPD, HF, recovering from a coronary artery disease related event, and taking diuretic medication).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Hospital, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Cohort | Pathologic Cohort
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Cohort | Pathologic Cohort | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 8 | 23
  >=65 years | 5 | 12 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 10 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.92 (3.47) | 33.73 (7.37) | 29.83 (5.42)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient for Accuracy of Test Device vs Reference Device
Description: Correlation Coefficient for Respiration Rate accuracy (test device vs reference device).
Time Frame: Device reading (3 minutes)
Population: Analysis of the Healthy Cohort for both Supine and Upright positions
Measure: Number; unit: Correlation Coefficient
Units Other Than Participants: Number of Measurements
Groups:
- Supine Position: This data group is comprised of device measurements from the Supine position of the Healthy Cohort.
  Noninterventional and noninvasive: The ADI At-Home CPM (Cardiopulmonary Management) System is intended for adults undergoing monitoring for cardiopulmonary conditions under the direction of a licensed medical professional to measure, record, and periodically transmit physiological data.
- Upright Position: This data group is comprised of device measurements from the Upright position of the Healthy Cohort.
  Noninterventional and noninvasive: The ADI At-Home CPM (Cardiopulmonary Management) System is intended for adults undergoing monitoring for cardiopulmonary conditions under the direction of a licensed medical professional to measure, record, and periodically transmit physiological data.
Arm/Group | Supine Position | Upright Position
Number analyzed (Participants) | 20 | 20
Number analyzed (Number of Measurements) | 150 | 133
Correlation Coefficient | 0.99 | 0.95

2. Primary Outcome: Root Mean Square Error Accuracy Between CPM and Reference Device for Respiration Rate
Time Frame: Device reading (3 minutes)
Population: Analysis of the Healthy Cohort for both Supine and Upright positions
Measure: Number; unit: Breaths per minute
Units Other Than Participants: Device measurements
Arm/Group | Supine Position | Upright Position
Number analyzed (Participants) | 20 | 20
Number analyzed (Device measurements) | 150 | 133
Breaths per minute | 1.74 | 3.26

3. Primary Outcome: Correlation Coefficient Between Reference Tidal Volume (TV) and Test Device Relative Tidal Volume (rTV)
Description: Accuracy of CPM System calculated rTV (relative Tidal Volume) as compared to reference device calculated TV (Tidal Volume)
Time Frame: Device reading (3 minutes)
Population: Analysis of Supine and Upright Positions for Healthy Cohort
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Units Other Than Participants: Device measurements
Groups:
- Upright Position: This data group is comprised of device measurements from the Supine position of the Healthy Cohort.
  Noninterventional and noninvasive: The ADI At-Home CPM (Cardiopulmonary Management) System is intended for adults undergoing monitoring for cardiopulmonary conditions under the direction of a licensed medical professional to measure, record, and periodically transmit physiological data.
Arm/Group | Supine Position | Upright Position
Number analyzed (Participants) | 20 | 20
Number analyzed (Device measurements) | 260 | 260
Correlation coefficient | 0.98 [0.96 to 0.99] | 0.94 [0.91 to 0.97]

4. Primary Outcome: Standard Deviation of Thoracic Impedance
Description: Analyses were performed to quantify replication variability. The analysis used Mixed models for repeated measures (MMRM) to obtain the variance component estimates controlling for changes in true status as measured by the bioimpedance reference. The variance components include replication variance within application with three measurements per application (i.e., short-term variance) and application variance with three applications, including an application one hour later (longer-term variance). The model also includes subject to subject variance (adjusted for changes in the bioimpedance reference). Variability among applications is partially explained by changes in bioimpedance reference. Total variance is partitioned into measurement variance, application variance, and subject variance.
Time Frame: device reading (3 minutes)
Measure: Number (95% Confidence Interval); unit: Ohms
Units Other Than Participants: device measurements
Arm/Group | Pathologic Cohort
Number analyzed (Participants) | 20
Number analyzed (device measurements) | 180
Ohms | 2.08 [1.84 to 2.38]

5. Primary Outcome: Magnitude of Drift for Thoracic Impedance
Description: The magnitude of drift was evaluated by comparing the magnitude of this longer-term variance to the short term (replication) variance in relative term and comparing the absolute incremental contribution of the longer-term standard deviation to 6 ohms. If adding application variance (controlling for change in bioimpedance reference) does not appreciably increase the total nonsubject variance, no appreciable drift across will have been demonstrated.
Time Frame: Device reading (3 minutes)
Measure: Number (95% Confidence Interval); unit: Ohms
Units Other Than Participants: device measurements
Arm/Group | Pathologic Cohort
Number analyzed (Participants) | 20
Number analyzed (device measurements) | 180
Ohms | 2.75 [2.46 to 3.13]

6. Secondary Outcome: ECG Heart Rate Confirmation
Description: Confirm that ECG characteristics align with those from bench results using a simulator
Time Frame: Device measurement (3 minutes)
Population: ECG Strips from Pathologic Cohort
Measure: Number; unit: Beats per minute (BPM)
Units Other Than Participants: Device measurement ECG Strips
Groups:
- Cardiologist 1; Cardiologist 2: Results when compared to metrics reported by Cardiologist 1 reading the ECG Strip
Arm/Group | Cardiologist 1 | Cardiologist 2
Number analyzed (Participants) | 20 | 20
Number analyzed (Device measurement ECG Strips) | 60 | 60
Beats per minute (BPM)
  Maximum Absolute Error | 17 | 15
  Mean Absolute Error | 4.93 | 5.5
  Bias Error | -4.67 | -5.07
  Standard Deviation of Error | 4.79 | 5.21
  Coefficient of determination | 0.91 | 0.90

7. Secondary Outcome: Skin Temperature Confirmation.
Description: Confirm that ECG characteristics align with those from bench results using a simulator
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees Celcius
Units Other Than Participants: device measurements
Arm/Group | Pathologic Cohort
Number analyzed (Participants) | 20
Number analyzed (device measurements) | 200
degrees Celcius | 26.33 (0.46)

8. Secondary Outcome: ECG Confirmation for Abnormal Rhythms
Description: Comparing device ECG Abnormal Rhythm Flags raised by CPM system to cardiologist atrial fibrillation annotation of device ECG strips (3 strips per participant). Counts determine total number of ECG strips flagged with abnormalities if the CPM device or cardiologist annotated atrial fibrillation.
Time Frame: Device measurement (3 minutes)
Population: ECG Strips from Pathologic Cohort
Measure: Number; unit: ECG Strips with atrial fibrillation
Units Other Than Participants: Device measurement ECG Strips
Groups:
- CPM Abnormal Rhythm Flag: CPM System Flag's for abnormal rhythm
- Cardiologist 1; Cardiologist 2: Cardiologist 2 annotation of CPM Device ECG strip for abnormal rhythms
Arm/Group | CPM Abnormal Rhythm Flag | Cardiologist 1 | Cardiologist 2
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Device measurement ECG Strips) | 60 | 60 | 60
ECG Strips with atrial fibrillation | 6 | 6 | 6

9. Secondary Outcome: ECG QRS, QT and QTc Confirmation
Description: Confirm that ECG characteristics align with those from bench results using a simulator
Time Frame: device reading (3 minutes)
Population: ECG Strips from Pathologic Cohort
Measure: Number; unit: ms (millisecond)
Units Other Than Participants: Device measurement ECG Strips
Arm/Group | Cardiologist 1 | Cardiologist 2
Number analyzed (Participants) | 20 | 20
Number analyzed (Device measurement ECG Strips) | 60 | 60
ms (millisecond)
  QRS width - Maximum Absolute Error | 57.5 | 57.5
  QRS Width - Mean Absolute Error | 26.4 | 27.4
  QRS Width - Bias Error | 25.4 | 26.3
  QRS Width - Standard Deviation of Error | 17.4 | 18.3
  QRS Width - Coefficient of determination | 0.48 | 0.45
  QT interval - Mean Absolute Error | 51.7 | 49.2
  QT interval - Bias Error | 24.9 | 22.6
  QT interval - Standard Deviation of Error | 66.9 | 67.2
  QT interval - Coefficient of determination | 0.22 | 0.21
  QTc interval - Maximum Absolute Error | 257.4 | 257.4
  QTc interval - Mean Absolute Error | 50.8 | 48.4
  QTc interval - Bias Error | 10.6 | 7.0
  QTc interval - Standard Deviation of Error | 77.8 | 77.0
  QTc interval - Coefficient of determination | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Healthy Cohort | Pathologic Cohort
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04865640/Prot_SAP_000.pdf